CLINICAL TRIAL: NCT03925727
Title: Multi-Center, Randomized,Double-Masked, Vehicle-Controlled Study to Assess the Safety and Efficacy Study of Tavilermide Ophthalmic Solutions for the Treatment of Dry Eye
Brief Title: Tavilermide Ophthalmic Solution for the Treatment of Dry Eye
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mimetogen Pharmaceuticals USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MIM-728
Record Dates: First submitted 2019-04-19; First posted 2019-04-24 (Actual); Results first posted 2023-03-09 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Keratoconjunctivitis Sicca; Dry Eye
MeSH Terms: conditions — Keratoconjunctivitis Sicca; Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 1% Tavilermide ophthalmic solution (Experimental)
  Interventions: Drug: Tavilermide ophthalmic solution
- 5% Tavilermide ophthalmic solution (Experimental)
  Interventions: Drug: Tavilermide ophthalmic solution
- Vehicle ophthalmic solution (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tavilermide ophthalmic solution — BID topical dosing
  Arms: 1% Tavilermide ophthalmic solution; 5% Tavilermide ophthalmic solution
Other: Placebo — BID topical dosing
  Arms: Vehicle ophthalmic solution

SUMMARY:
The purpose of this study is to assess the safety and efficacy of 5% tavilermide and 1% tavilermide ophthalmic solutions compared with placebo ophthalmic solution in treating the signs and symptoms of dry eye.

ELIGIBILITY:
Inclusion Criteria:

* Subject-reported history of dry eye disease in both eyes for at least 6 months;
* History of use of artificial tear eye drops for dry eye symptoms;
* Total score of ≥40 on SANDE;
* TFBUT;
* Corneal fluorescein staining;
* Lissamine green conjunctival staining;
* Schirmer's test score.

Exclusion Criteria:

* Have participated in a previous tavilermide (MIM-D3) study;
* Have clinically significant slit lamp findings at Visit 1;
* Have a history of lacrimal duct obstruction within 12 months of Visit 1;
* Have an uncontrolled systemic disease;
* Be a woman who is pregnant, nursing or planning a pregnancy;
* Be a woman of childbearing potential who is not using an acceptable means of birth control;
* Have a condition or be in a situation which the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study;
* Be currently enrolled in an investigational drug or device study or have used an investigational drug or device within 45 days prior to Visit 1.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 623 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2020-06-11 (Actual); Study Completion 2020-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Meerovitch, PhD, Study Director — Mimetogen Pharmaceuticals
Locations (22):
- United States (22):
  - Tavilermide Investigational Site, Phoenix, Arizona
  - Tavilermide Investigational Site, Los Angeles, California
  - Tavilermide Investigational Site, Newport Beach, California
  - Tavilermide Investigational Site, Fort Collins, Colorado
  - Tavilermide Investigational Site, Littleton, Colorado
  - Tavilermide Investigational Site, Boynton Beach, Florida
  - Tavilermide Investigational Site, Bradenton, Florida
  - Tavilermide Investigational Site, Coral Springs, Florida
  - Tavilermide Investigational Site, Ocala, Florida
  - Tavilermide Investigational Site, Indianapolis, Indiana
  - Tavilermide Investigational Site, Sioux City, Iowa
  - Tavilermide Investigational Site, Lexington, Kentucky
  - Tavilermide Investigational Site, Louisville, Kentucky
  - Tavilermide Investigational Site, St Louis, Missouri
  - Tavilermide Investigational Site, Shelby, North Carolina
  - Tavilermide Investigational Site, Cincinnati, Ohio
  - Tavilermide Investigational Site, Mason, Ohio
  - Tavilermide Investigational Site, Rapid City, South Dakota
  - Tavilermide Investigational Site, Maryville, Tennessee
  - Tavilermide Investigational Site, Nashville, Tennessee
  - Tavilermide Investigational Site, San Antonio, Texas
  - Tavilermide Investigational Site, Kenosha, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Tavilermide 5%; Tavilermide 1%: Twice daily topical ocular dosing for 12 weeks
- Placebo: Twice daily topical ocular dosing for 12 weeks (vehicle)
Period: Overall Study
Arm/Group | Tavilermide 5% | Tavilermide 1% | Placebo
Started | 263 | 100 | 260
Completed | 244 | 94 | 242
Not Completed | 19 | 6 | 18
Not completed — Adverse Event | 4 | 0 | 3
Not completed — Protocol Violation | 1 | 2 | 2
Not completed — Withdrawal by Subject | 3 | 2 | 4
Not completed — Administrative Reasons | 3 | 1 | 2
Not completed — Randomized in error or Disqualified | 8 | 1 | 7

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) set included all randomized participants
Groups:
- Tavilermide 5%; Tavilermide 1%: Tavilermide ophthalmic solution: BID topical dosing
- Vehicle: Placebo: BID topical dosing
- Total: Total of all reporting groups
Arm/Group | Tavilermide 5% | Tavilermide 1% | Vehicle | Total
Number analyzed (Participants) | 257 | 97 | 253 | 607
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.1 (13.47) | 59.7 (14.63) | 60.5 (14.00) | 60.6 (13.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 201 | 80 | 184 | 465
  Male | 56 | 17 | 69 | 142
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 9 | 29 | 63
  Not Hispanic or Latino | 232 | 88 | 224 | 544
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 2 | 7
  Asian | 11 | 5 | 8 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 21 | 8 | 27 | 56
  White | 219 | 81 | 213 | 513
  More than one race | 0 | 1 | 2 | 3
  Unknown or Not Reported | 3 | 0 | 1 | 4
Eye Dryness Score [Mean (Standard Deviation); unit: units on a scale] — Visual Analog Scale (0 to 100 Scale, Higher is Worse)
  units on a scale | 63.3 (20.38) | 65.8 (19.06) | 65.0 (20.22) | 64.4 (20.10)
Total Corneal Fluorescein Staining [Mean (Standard Deviation); unit: units on a scale] — National Eye Institute Scale (0 to 15, Higher is Worse)
  units on a scale | 7.4 (1.92) | 7.4 (1.77) | 7.6 (2.06) | 7.5 (1.96)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Eye Dryness Score as Measured by the VAS
Description: The Visual Analog Scale (VAS) where subjects were asked to rate their eye dryness (OU) by placing a vertical mark on the horizontal line to indicate their current level of discomfort. 0 mm corresponds to "No Discomfort," and 100 mm corresponds to "Maximal Discomfort." The length of the assessment line is 100 mm.
Time Frame: Baseline to Day 85 in 5% Tavilermide versus Placebo
Population: ITT Population with Markov Chain Monte Carlo (MCMC) on all randomized subjects
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Tavilermide 5%; Tavilermide 1%: BID topical ocular dosing
- Placebo: BID topical dosing (vehicle)
Arm/Group | Tavilermide 5% | Tavilermide 1% | Placebo
Number analyzed (Participants) | 257 | 97 | 253
score on a scale | -15.1 (1.64) | -20.6 (2.66) | -16.5 (1.67)
Statistical Analysis 1: Comparison: Tavilermide 5% vs Placebo; Test type: Superiority; p = 0.5533, ANCOVA; Mean Difference (Net) = 1.4, 95% CI 2-sided [-3.2 to 6]

2. Primary Outcome: Change From Baseline in Total Corneal Fluorescein Staining as Measured by the NEI Scale
Description: The National Eye Institute (NEI) scale is a standardized grading system of 0-3 was used for each of the 5 areas on each cornea (central, superior, temporal, nasal, and inferior) . Grade 0 was specified when no staining is present. The maximum score was 15. Study eye is the 'worse eye', defined as the eye with worse (higher) score at baseline.
Time Frame: Baseline to Day 85 in 5% Tavilermide versus Placebo
Population: ITT Population with MCMC on all randomized subjects
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Tavilermide 5%; Tavilermide 1%: BID topical dosing
Arm/Group | Tavilermide 5% | Tavilermide 1% | Placebo
Number analyzed (Participants) | 257 | 97 | 253
units on a scale | -2.6 (0.17) | -2.3 (0.28) | -2.1 (0.17)
Statistical Analysis 1: Comparison: Tavilermide 5% vs Placebo; Test type: Superiority; p = 0.0192, ANCOVA; Mean Difference (Net) = -0.6, 95% CI 2-sided [-1.1 to -0.1]

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Adverse event collection was on the safety population which included all randomized subjects who received at least one dose of the investigational product.
Groups:
- Tavilermide 5%; Tavilermide 1%: Twice daily topical dosing
- Placebo: Twice daily topical dosing (vehicle)
Arm/Group | Tavilermide 5% | Tavilermide 1% | Placebo
All-Cause Mortality (participants affected / at risk) | 1/261 | 0/99 | 0/255
Serious Adverse Events (participants affected / at risk) | 2/261 | 0/99 | 3/255
Other Adverse Events (participants affected / at risk) | 16/261 | 1/99 | 8/255
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tavilermide 5% (N=261) | Tavilermide 1% (N=99) | Placebo (N=255)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tavilermide 5% (N=261) | Tavilermide 1% (N=99) | Placebo (N=255)
Instillation site pain (General disorders) | 16 (25) | 1 (1) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor, or its designee, shall have the right to coordinate one or more publications of the aggregate multi-site Study results. Accordingly, Investigator agrees not to publish or present the results of the Study until such time as the aggregate multi-site Study results are published.

DOCUMENTS (2):
  • Study Protocol (2019-07-03): https://cdn.clinicaltrials.gov/large-docs/27/NCT03925727/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-15): https://cdn.clinicaltrials.gov/large-docs/27/NCT03925727/SAP_001.pdf